CLINICAL TRIAL: NCT03193970
Title: Measuring Surgical Recovery After Radical Cystectomy
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA15-0026; NCI-2018-01433 (Registry Identifier: NCI CTRP-Clinical Trials Registry)
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Registry; Post-surgical outcomes; Radical cystectomy; MD Anderson Symptom inventory; MDASI
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder Cancer Patients Undergoing Radical Cystectomy: Prospective registry of bladder cancer patients undergoing radical cystectomy at MD Anderson Cancer Center and the collaborating centers.
  Interventions: Behavioral: Post-Operative Recovery Registry

INTERVENTIONS:
Behavioral: Post-Operative Recovery Registry — Multi-institutional prospective database of patients with bladder cancer undergoing radical cystectomy.

SUMMARY:
The intent of this study is to establish a registry of post-surgical outcomes in patients undergoing radical cystectomy at MD Anderson Cancer Center and the collaborating institutions. The goals of this initiative are to obtain a detailed baseline of multiple patient-reported outcomes (PRO) and clinician-reported outcomes (CRO) as well as various presenting conditions associated with them, so that future quality improvement interventions can be evaluated accurately as to their relative contribution to improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Bladder cancer patients undergoing radical cystectomy at the MD Anderson Cancer Center and the collaborating centers.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients undergoing radical cystectomy at the MD Anderson Cancer Center and the collaborating centers.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-04-30 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Surgical Outcomes in Patients Undergoing Radical Cystectomy | 3 months
  Post-surgical outcomes determined from patient-reported assessment of symptom burden using the MD Anderson Symptom Inventory (MDASI-BLC form).

CONTACTS AND LOCATIONS:
Overall Officials: Neema Navai, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (11):
- United States (11):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Lawrence, Kansas
  - John Hopkins Medical Institutions, Baltimore, Maryland
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Winthrop University Hospital, Mineola, New York
  - University of Rochester, Rochester, New York
  - University of Texas - Southwestern, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org